CLINICAL TRIAL: NCT04425096
Title: The Effect of Skin to Skin Contact on Postpartum Hemorrhage, Pain And Breastfeeding: Randomized Controlled Trial
Brief Title: The Effect of Skin to Skin Contact on Postpartum Hemorrhage, Pain And Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Associate Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018/066
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Skin to Skin Contact
Keywords: Postpartum Pain; Breastfeeding; Beta Endorphin; Oxytocin; Postpartum Hemorrhage; Skin to Skin Contact
MeSH Terms: conditions — Breast Feeding; Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: Randomized controlled single-blind experimental study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin to skin contact (Experimental): The mothers and their babies in the experimental group received a 30-minute skin to skin contact immediately after birth (n:34)
  Interventions: Other: Skin to skin contact
- Routine care (No Intervention): The babies in the control group received routine care (n:34)

INTERVENTIONS:
Other: Skin to skin contact — Skin to skin contact
  Arms: Skin to skin contact

SUMMARY:
The aim of this study was to determine the effect of postpartum hemorrhage, pain and onset of early breastfeeding so that the skin applied at the third stage of birth is in contact with the skin. Material and Method: The study was carried out as a randomized controlled single-blind experimental study. The sample consists of 68 healthy mother and baby pairs. Skin contact with mothers and babies in the experimental group will be applied for 34 minutes immediately after birth. Routine care will be applied to the babies in the control group. Data will be collected using Personal Information Form, Visual Analogue Scale, LATCH Breastfeeding Diagnostic Scale, Breastfeeding Self-Efficacy Scale, postpartum hemorrhage follow-up bag, pad and oxytocin, ᵦ endorphine analysis results.

were collected using Personal Information Form, Visual Analogue Scale, LATCH Breastfeeding Diagnostic Scale, Breastfeeding Self-Efficacy Scale, postpartum bleeding follow-up bag, pad and oxytocin, ᵦ endorphin analysis results.

DETAILED DESCRIPTION:
Implementation of the Practice of the Study; In the standard practice of the delivery room clinic, where the study was planned, babies are clamped as soon as they are born, and their routine care (such as K vit and hepatitis B vaccine application) is taken under the radiant heater. The skin contact can not be applied between the baby and the mother. After the baby is cared, until the mother is transferred to the postpartum clinic, the baby is wrapped in a clean cotton sterile cloth under a radiant heater in the baby room.

Routine care was applied to the babies of the control group mothers. No physical contact with the babies of the control group mothers was performed, standard applications were applied in the clinic (placing the baby under the radiant heater for clamping the umbilical cord as soon as it was born, K-vit application, Hepatitis B vaccine application etc.).

As soon as the babies of the mothers in the experimental group were born, the babies were placed in a prone position with skin contact on their mothers' bare belly. The baby was gently dried, covered with a blanket and a beret was worn. The umbilical cord of the baby was clamped late (approximately 1-3 minutes). The baby was kept in this position for 30 minutes and then taken under the radiant heater for routine care.

Blood was collected from women in the experimental and control groups for the 1st and 30th minutes after the birth of the baby for oxytocin and ᵦ endorphin analysis. After for both groups, VAS was applied after 2nd and 6th hours after birth, LATCH Breastfeeding Assessment and BSS were applied in 24th hour and 1 week later of the birth. Immediately after birth, a postpartum hemorrhage follow-up bag was placed on the gynecological table and followed by a bleeding bag until the mother got up from the gynecological table. When women were taken to bed from gynecological table, bleeding was followed up with a perineal pad. Weights of pad and mattress protections of women were weighed at 24 hours because normal women were discharged at 24 hours after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-35 years,
* having a single pregnancy,
* literate,
* between 37-42 gestational week,
* hemoglobin level of 10 g and above,
* without chronic, mental and psychological disease

Infants;

* without congenital anomalies,
* with a first Apgar score of 8 and above,
* birth weight between 2500 - 4000 g
* no obstruction to oral feeding

Exclusion Criteria:

* Induction practice,
* multiparity,
* any risky condition development in the mother and baby during or after birth

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Oxytocin Analysis | 1 minute -30 minutes.
  Oxytocin 1minute level
ᵦ endorphin Analysis | 1 minute -30 minutes.
  ᵦ endorphin 1 minute
VAS (Visuel Analog Scale) | 2nd hour- 6 th hour
  VAS is a commonly used measurement tool for determining the degree of pain. The patient is asked to mark his or her pain on a 10 cm ruler that writes painlessness (0) on one end and the most severe pain (10) on the other end
LATCH Breastfeeding Assessment Tool | 24th hour -1st week
  LATCH (L: is for how well the infantlatches onto the breast, A: is for the amount of audibleswallowing noted, T: is for the mother's nipple type/condition, C: is for the mother's level of comfort, and H: isfor the amount of help the mother needs to hold her infant tothe breast) assessment tool is based on observations and descriptions of effective breastfeeding, evaluates five characteristics of breastfeeding .The total score ranges from 0 to 10, with the higherscore representing successful breastfeeding.
Breastfeeding Self-Efficacy Scale | 24th hour -1st week
  Breastfeeding Self-Efficacy Scale; The 5-point Likert type scale consists of 14 items. Minimum 14 points, maximum 70 points can be obtained, and high scores indicate that breastfeeding selfefficacy is higher.
Postpartum Blood Bag | 24th hour
  Immediately after birth, a postpartum hemorrhage follow-up bag was placed on the gynecological table and followed by a bleeding bag until the mother got up from the gynecological table.
Total Postpartum Blood Loss | 24th hour
  Total Postpartum Blood Loss(postpartum blood bag +pad test ): Immediately after birth, a postpartum hemorrhage follow-up bag was placed on the gynecological table and followed by a bleeding bag until the mother got up from the gynecological table. When women were taken to bed from gynecological table, bleeding was followed up with a perineal pad. Weights of pad and mattress protections of women were weighed at 24 hours because normal women were discharged at 24 hours after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin AYDIN KARTAL, PhD, Study Director — Saglık Bilimleri U
Locations (1):
- Saglık Bilimleri Universitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alus Tokat, M. & Okumuş, H. (2013). The Effect of Antenatal Training Based on Strengthening the Perception of Breastfeeding Self-Efficacy on the Perception of Breastfeeding Self- Efficacy and Breastfeeding. Journal of Nursing Education and Research, 10, 21-29
- [Background] Annagür, B. & Annagür, A. (2012). Relationship of Postpartum Mental Status with Breastfeeding. Current Approaches in Psychiatry, 4, 279-292
- [Background] Çalısır, H., Karaçam, Z., Akgül, F.A. & Kurnaz, D.A. (2009). Validity and Reliability of the Turkish Form of the Postpartum Parenting Behavior Scale. Journal of Atatürk University School of Nursing, 12, 1-8
- [Background] Cong X, Ludington-Hoe SM, Hussain N, Cusson RM, Walsh S, Vazquez V, Briere CE, Vittner D. Parental oxytocin responses during skin-to-skin contact in pre-term infants. Early Hum Dev. 2015 Jul;91(7):401-6. doi: 10.1016/j.earlhumdev.2015.04.012. Epub 2015 May 16. PMID 25988992
- [Background] Cooijmans KHM, Beijers R, Rovers AC, de Weerth C. Effectiveness of skin-to-skin contact versus care-as-usual in mothers and their full-term infants: study protocol for a parallel-group randomized controlled trial. BMC Pediatr. 2017 Jul 6;17(1):154. doi: 10.1186/s12887-017-0906-9. PMID 28683833
- [Background] Edwards HM. Aetiology and treatment of severe postpartum haemorrhage. Dan Med J. 2018 Mar;65(3):B5444. PMID 29510809
- [Background] Essa R.M., İsmail N. & İsmail A. (2015). Effect of Early Maternal/Newborn Skin-To- Skin Contact After Birth On The Duration Of Third Stage Of Labor And İnitiation Of Breastfeeding. Journal of Nursing Education and Practice, 54, 98-107.
- [Background] Hughes KN, Rodriguez-Carter J, Hill J, Miller D, Gomez C. Using Skin-to-Skin Contact to Increase Exclusive Breastfeeding at a Military Medical Center. Nurs Womens Health. 2015 Dec-2016 Jan;19(6):478-89. doi: 10.1111/1751-486X.12244. PMID 26682656
- [Background] Karimi, A., Tara, F., Khadivzadeh, T. & Aghamohammadian, Sharbaf, H.R. (2013). The Effect of Skin to Skin Contact Immediately after Delivery on the Maternal Attachment and Anxiety Regarding Infant. Iran J Obstet Gynecol Infertil, 16, 7-15.
- [Background] Karimi, F.Z., Bagheri, S., Tara, F., Khadivzadeh, T. & Mousavi, Bazaz, S.M. (2014). Effect ofKangaroo Mother Care on breastfeeding self efficacy in primiparous women, 3 month after child birth. Iran J Obstet Gynecol Infertil, 17, 1-8.
- [Background] Linares AM, Wambach K, Rayens MK, Wiggins A, Coleman E, Dignan MB. Modeling the Influence of Early Skin-to-Skin Contact on Exclusive Breastfeeding in a Sample of Hispanic Immigrant Women. J Immigr Minor Health. 2017 Oct;19(5):1027-1034. doi: 10.1007/s10903-016-0380-8. PMID 26969615